CLINICAL TRIAL: NCT01358513
Title: An Observational PET/CT Study Examining the Role of Active Valvular Calcification and Inflammation in Patients With Aortic Stenosis
Brief Title: Role of Active Valvular Calcification and Inflammation in Patients With Aortic Stenosis
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: RING OF FIRE
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2015-01

CONDITIONS: Aortic Stenosis
Keywords: Positron Emission Tomography; Inflammation; Calcification
MeSH Terms: conditions — Aortic Valve Stenosis; Inflammation; Calcinosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In patients undergoing aortic valve replacement during the course of the trial we will retain samples of their aortic valve for histological studies.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Control Patients: Patients with normal aortic valves
- Aortic sclerosis: To undergo PET imaging and follow up with CT and echo for 2 years
- Mild Aortic stenosis: To undergo PET imaging and follow up with CT and echo for 2 years
- Moderate Aortic stenosis: To undergo PET imaging and follow up with CT and echo for 2 years
- Severe aortic stenosis: To undergo PET imaging and follow up with CT and echo for 2 years

SUMMARY:
The aortic valve is the main outlet valve from the heart. This valve can become diseased and narrowed when it needs to be replaced with an artificial valve. Currently, this is the commonest reason for someone to undergo a heart valve operation in the UK. Unfortunately, there are no medical treatments that can prevent or delay the progression of this disease process. Here, the investigators propose to use new state-of-the-art imaging techniques to better understand the disease process so that the investigators can effectively design and assess potential new treatments. The ultimate aim is to stop this disease before patients need to have surgery. In addition the investigators believe this technique will allow us to predict the rate of progression of the disease

DETAILED DESCRIPTION:
Aortic stenosis is the commonest valvular heart disease in the western world and is the leading indication for valve surgery. Histological studies have suggested similarities with atherosclerosis including inflammation, lipid deposition, increased macrophage activity and calcification. However, recent randomised controlled trials have failed to demonstrate a reduction in the rate of disease progression with statin therapy and the investigators believe there is now a need to re-evaluate the underlying factors involved in the initiation and progression of aortic stenosis. The investigators propose to assess the role of inflammation and calcification in the pathogenesis and progression of aortic stenosis by using positron emission tomography with [18F]-fluorodeoxyglucose and [18F-]-fluoride in patients with a range of aortic valve disease. The investigators hypothesise that increasing severity of valvular inflammation and calcification will correlate with disease severity and rate of disease progression. This work will lay the foundation for the subsequent application of interventions targeted at inflammation and calcification.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years

Exclusion Criteria:

* Age < 50 years
* Life expectancy < 2 years
* Insulin dependent diabetes mellitus
* Connective Tissue disorders

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit 168 patients: 24 control patients, 24 mild, 48 moderate and 48 severe aortic stenosis
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2010-07; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Aortic Valve Peak Velocity | 2 years
  We beleive NaF and FDG uptake in the valve will predict rate of progression of the disease. Disease severity will be measured by the aortic valve peak velocity

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Cardiovascular Sciences, University of Edinburgh, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Derived] Fletcher AJ, Tew YY, Tzolos E, Joshi SS, Kaczynski J, Nash J, Debono S, Lembo M, Kwiecinski J, Bing R, Syed MBJ, Doris MK, van Beek EJR, Moss AJ, Jenkins WS, Walker NL, Joshi NV, Pawade TA, Adamson PD, Whiteley WN, Wardlaw JM, Slomka PJ, Williams MC, Newby DE, Dweck MR. Thoracic Aortic 18F-Sodium Fluoride Activity and Ischemic Stroke in Patients With Established Cardiovascular Disease. JACC Cardiovasc Imaging. 2022 Jul;15(7):1274-1288. doi: 10.1016/j.jcmg.2021.12.013. Epub 2022 Feb 16. PMID 35183477
- [Derived] Pawade T, Clavel MA, Tribouilloy C, Dreyfus J, Mathieu T, Tastet L, Renard C, Gun M, Jenkins WSA, Macron L, Sechrist JW, Lacomis JM, Nguyen V, Galian Gay L, Cuellar Calabria H, Ntalas I, Cartlidge TRG, Prendergast B, Rajani R, Evangelista A, Cavalcante JL, Newby DE, Pibarot P, Messika Zeitoun D, Dweck MR. Computed Tomography Aortic Valve Calcium Scoring in Patients With Aortic Stenosis. Circ Cardiovasc Imaging. 2018 Mar;11(3):e007146. doi: 10.1161/CIRCIMAGING.117.007146. PMID 29555836
- [Derived] Dweck MR, Jenkins WS, Vesey AT, Pringle MA, Chin CW, Malley TS, Cowie WJ, Tsampasian V, Richardson H, Fletcher A, Wallace WA, Pessotto R, van Beek EJ, Boon NA, Rudd JH, Newby DE. 18F-sodium fluoride uptake is a marker of active calcification and disease progression in patients with aortic stenosis. Circ Cardiovasc Imaging. 2014 Mar;7(2):371-8. doi: 10.1161/CIRCIMAGING.113.001508. Epub 2014 Feb 7. PMID 24508669
- [Derived] Dweck MR, Khaw HJ, Sng GK, Luo EL, Baird A, Williams MC, Makiello P, Mirsadraee S, Joshi NV, van Beek EJ, Boon NA, Rudd JH, Newby DE. Aortic stenosis, atherosclerosis, and skeletal bone: is there a common link with calcification and inflammation? Eur Heart J. 2013 Jun;34(21):1567-74. doi: 10.1093/eurheartj/eht034. Epub 2013 Feb 7. PMID 23391586
- [Derived] Dweck MR, Chow MW, Joshi NV, Williams MC, Jones C, Fletcher AM, Richardson H, White A, McKillop G, van Beek EJ, Boon NA, Rudd JH, Newby DE. Coronary arterial 18F-sodium fluoride uptake: a novel marker of plaque biology. J Am Coll Cardiol. 2012 Apr 24;59(17):1539-48. doi: 10.1016/j.jacc.2011.12.037. PMID 22516444
- [Derived] Dweck MR, Jones C, Joshi NV, Fletcher AM, Richardson H, White A, Marsden M, Pessotto R, Clark JC, Wallace WA, Salter DM, McKillop G, van Beek EJ, Boon NA, Rudd JH, Newby DE. Assessment of valvular calcification and inflammation by positron emission tomography in patients with aortic stenosis. Circulation. 2012 Jan 3;125(1):76-86. doi: 10.1161/CIRCULATIONAHA.111.051052. Epub 2011 Nov 16. PMID 22090163